CLINICAL TRIAL: NCT01763996
Title: The Influence of Febuxostat on Coronary Artery Endothelial Dysfunction in Subjects With Chronic Stable Angina: A Phase 4 Randomized, Placebo-Controlled, Double-Blind, Cross-Over Study
Brief Title: The Influence of Febuxostat on Coronary Artery Endothelial Dysfunction in Participants With Chronic Stable Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CCR-FEB-002; U1111-1136-2270 (Registry Identifier: WHO)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: Drug therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: Febuxostat 80 mg + Placebo (Experimental): Febuxostat 80 mg, capsules, orally, once daily for 6 weeks in Period 1, followed by febuxostat placebo-matching capsules, orally, once daily for up to 6 weeks in Period 2.
  Interventions: Drug: Febuxostat; Drug: Febuxostat placebo
- Sequence 2: Placebo + Febuxostat 80 mg (Experimental): Febuxostat placebo-matching capsules, orally, once daily for 6 weeks in Period 1, followed by febuxostat 80 mg, capsules, orally, once daily for up to 6 weeks in Period 2.
  Interventions: Drug: Febuxostat; Drug: Febuxostat placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat capsules
Drug: Febuxostat placebo — Febuxostat placebo-matching capsules

SUMMARY:
The purpose of this study is to assess the effect of febuxostat on coronary artery flow in patients with coronary artery disease.

DETAILED DESCRIPTION:
The drug being tested in this study is called febuxostat. Febuxostat is being tested to treat people who have angina. This study will look at the heart and blood flow of people who take febuxostat.

The study will enroll approximately 30 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups (or sequences)-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Sequence 1: 6 weeks febuxostat followed by 6 weeks of placebo.
* Sequence 2: 6 week placebo followed by 6 weeks of febuxostat

All participants will be asked to take one capsule at the same time each day throughout the study. All participants will be asked to record any time they have angina symptoms during the study.

This single-center trial will be conducted in the United States. The overall time to participate in this study is 16 weeks. Participants will make 7 visits to the clinic including a final visit 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a serum urate ≥4.0 mg/dL.
4. Has a history of coronary artery disease, defined as:

   1. ≥50 % stenosis of ≥1 major coronary artery confirmed by angiography; OR
   2. Documented prior myocardial infarction (MI) by enzymes/electrocardiogram (ECG) changes; OR
   3. Documented prior exercise or pharmacologic stress/echo myocardial imaging study positive for ischemia.
5. Has estimated glomerular filtration rate (eGFR) ≥30 mL/min by Modification of Diet in Renal Disease (MDRD) at the screening visit.
6. Has a change in coronary artery flow from rest to isometric handgrip exercise of less than + 10 mL/min.
7. Is male or female and aged 18 to 85 years, inclusive.
8. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
9. Is on stable (30 days prior to Screening Day-21) medication doses prescribed for any underlying medical condition (ie, hypertension, angina) and is expected to remain on stable doses throughout the study duration.
10. Is able to take nitroglycerin for anginal symptoms during study procedures.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received allopurinol or febuxostat in a previous clinical study or as a therapeutic agent with-in 6 months of randomization.
3. Has gout or secondary hyperuricemia (eg, due to myeloproliferative disorder, or organ transplant) or has experienced a gout flare.
4. Has a history of xanthinuria.
5. Has known contraindication to magnetic resonance imaging (MRI) scanning
6. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
7. Has a history of hypersensitivity or allergies to febuxostat or nitroglycerin.
8. Has hemoglobin <10 g/L at Screening.
9. Has a history or clinical manifestations of a significant medical condition that might affect his/her ability to complete the study.
10. Has any of the following during Screening:

    1. New York Heart Association Class III or IV heart failure.
    2. Acute coronary syndrome or a coronary revascularization procedure within 2 months of Screening.
    3. Wolff-Parkinson-White syndrome.
    4. Pacemaker or implantable cardioverter defibrillator.
    5. Arrhythmias (ie, supraventricular tachycardia (SVT), atrial fibrillation/flutter, or ventricular tachycardia (VT) during Screening).
11. Has a recent history (within the last 2 months prior to Screening) of acute coronary syndrome or a coronary revascularization procedure, MI, heart failure, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
12. Has a contraindication for using nitrates (severe anemia, increased intracranial pressure, and those with a known sensitivity or hypersensitivity to nitroglycerin or its ingredients, or other nitrates or nitrites; concomitant use either regularly and/or intermittently, with phosphodiesterase type 5 (PDE5) inhibitors).
13. Has unstable angina that:

    1. Occurs when the patient is at rest.
    2. Is prolonged, usually greater than 20 minutes.
    3. Occurs with increasing in intensity, duration, and/or frequency.
    4. Responds poorly to nitroglycerin (ie, does not go away after three doses of nitroglycerin or returns after the nitroglycerin helped at first).
14. Is unable to exercise sufficiently to complete exercise treadmill test (ETT) due to leg claudication, arthritis, deconditioning, or associated pulmonary disease.
15. Has severe or critical valvular disease documented by echocardiogram, or congenital heart disease.
16. The subject has left ventricular ejection fraction (LVEF) less than 35%, as documented by echocardiogram, left ventriculogram, or gated blood pool scan..
17. The subject has clinically significant cardiac conduction defects (ie, second- or third-degree atrioventricular block, or sick sinus syndrome) at Screening
18. Has hypertrophic cardiomyopathy.
19. Has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level of greater than 2.0 times the upper limit of normal, has active liver disease, or jaundice.
20. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the Screening Visit.
21. Is required or expected to require excluded medications including digoxin or digoxin-containing compounds.
22. If female, is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
23. Has participated in another clinical trial within the past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- [Derived] Hays AG, Iantorno M, Schar M, Lai S, Czarny M, Breton E, Palmer RN, Whelton A, Weiss RG, Gerstenblith G. The influence of febuxostat on coronary artery endothelial dysfunction in patients with coronary artery disease: A phase 4 randomized, placebo-controlled, double-blind, crossover trial. Am Heart J. 2018 Mar;197:85-93. doi: 10.1016/j.ahj.2017.11.006. Epub 2017 Nov 23. PMID 29447788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United States from 29 May 2013 (first participant signed the formed consent form) to 14 April 2015.
Pre-assignment Details: Participants with a diagnosis of chronic stable angina were enrolled in one of 2 sequence cross-over arms: (1) febuxostat 80 mg for 6 weeks then placebo for 6 weeks, or (2) placebo for 6 weeks then febuxostat 80 mg for 6 weeks.
Period: Treatment Period 1
Arm/Group | Sequence 1: Febuxostat 80 mg + Placebo | Sequence 2: Placebo + Febuxostat 80 mg
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: Febuxostat 80 mg + Placebo | Sequence 2: Placebo + Febuxostat 80 mg
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- All Participants: All participants who were randomized and received study drug (febuxostat 80 mg and placebo) during the study.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 5
  White | 25
Region of Enrollment [Number; unit: participants]
  United States | 30
Height [Mean (Standard Deviation); unit: cm] | 176 (7.7)
Weight [Mean (Standard Deviation); unit: kg] | 87.8 (16)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (4.12)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent] | 56.8 (9.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Coronary Artery Flow From Rest to Isometric Handgrip (IHG) Exercise at the End of the Administration of Febuxostat and Placebo
Description: Coronary artery flow was measured using magnetic resonance imaging (MRI) at rest and during sustained isometric (static) handgrip exercises. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Groups:
- Placebo: Febuxostat placebo-matching capsules, orally, once daily for up to 6 weeks in Period 1 or 2.
- Febuxostat 80 mg: Febuxostat 80 mg, capsules, orally, once daily for up to 6 weeks in Period 1 or 2.
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 29 | 29
mL/min | 8.8 [0.40 to 17.28] | 10.7 [2.23 to 19.11]
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 80 mg; Test type: Superiority or Other; p = 0.756, ANOVA — 0.05 level of significance; Analysis of variance (ANOVA) model that includes sequence, period, and treatment as fixed factors and subjects within sequence as a random factor; LS Mean Difference = 1.8, 95% CI 2-sided [-10.10 to 13.76]

2. Secondary Outcome: Change in Coronary Artery Cross-Sectional Area From Rest to IHG Exercise at the End of the Administration of Febuxostat and Placebo
Description: Coronary artery cross-sectional area was measured by MRI at rest and during sustained isometric (static) handgrip exercise. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 29 | 29
mm^2 | 0.45 [-0.177 to 1.074] | 0.03 [-0.595 to 0.656]

3. Secondary Outcome: Change in Coronary Flow Velocity From Rest to IHG Exercise at the End of the Administration of Febuxostat and Placebo
Description: Coronary flow velocity was measured by MRI at rest and during sustained isometric (static) handgrip exercise. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/second
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 29 | 29
cm/second | 1.6 [-0.10 to 3.40] | 2.2 [0.43 to 3.93]

4. Secondary Outcome: Change in Coronary Artery Flow Following the Administration of Sublingual Nitroglycerin at the End of the Administration of Febuxostat and Placebo
Description: Coronary artery flow was measured by MRI before and following administration of nitroglycerin under the tongue. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, who used nitroglycerin.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 11 | 15
mL/min | 17.0 [-6.00 to 39.98] | 13.0 [-2.53 to 28.43]

5. Secondary Outcome: Change in Coronary Artery Cross Sectional Area Following the Administration of Sublingual Nitroglycerin at the End of the Administration of Febuxostat and Placebo
Description: Coronary artery cross sectional area was measured by MRI before and following administration of nitroglycerin under the tongue. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 11 | 15
mm^2 | 3.35 [1.449 to 5.244] | 2.86 [1.582 to 4.138]

6. Secondary Outcome: Change in Coronary Flow Velocity Following the Administration of Sublingual Nitroglycerin at the End of the Administration of Febuxostat and Placebo
Description: Coronary flow velocity was measured by MRI before and following administration of nitroglycerin under the tongue. Data at the end of each treatment period was combined for the febuxostat and the placebo arms. A positive change from Baseline indicates improvement.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/second
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 11 | 15
cm/second | -0.95 [-4.120 to 2.213] | -0.66 [-2.792 to 1.472]

7. Secondary Outcome: Change in Time to Onset of ≥1 mm ST-Segment Depression During Exercise Treadmill Test (ETT)
Description: Time in seconds to ischemic ECG changes during ETT. Continuous electrocardiography (ECG) was performed during an exercise treadmill test (modified Bruce protocol) to assess the onset of ST-segment depression after administration of febuxostat or placebo for 6 weeks in participants with a normal ST segment at randomization. . Data at the end of each treatment period was combined for the febuxostat and the placebo arms.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with ischemic ECG changes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 4 | 2
seconds | 514 (252) | 316 (122)

8. Secondary Outcome: Change in Maximum ST-segment Depression During Exercise Treadmill Test
Description: Continuous ECG was performed during an exercise treadmill test (modified Bruce protocol) to assess the maximum ST-segment depression after 6 weeks of febuxostat or placebo treatment in participants with a normal ST segment at randomization. A negative change from Baseline indicates improvement. Data at the end of each treatment period was combined for the febuxostat and the placebo arms.
Time Frame: Baseline and at the end of each 6 week treatment period (Week 6 and Week 12)
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with ST segment change.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 4 | 2
mm | 1.3 (0.5) | 1.5 (0.7)

9. Secondary Outcome: Percentage of Participants Stopping Exercise Treadmill Test Due to Angina at the End of the Administration of Febuxostat and Placebo
Description: An exercise treadmill test (modified Bruce protocol) was performed. Data at the end of each treatment period was combined for the febuxostat and the placebo arms.
Time Frame: At the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 30 | 28
percentage of participants | 0.0 | 3.6

10. Secondary Outcome: Time to Onset of Angina During Exercise Treadmill Test at the End of the Administration of Febuxostat and Placebo
Description: Time in seconds to ischemic chest pain/ angina during ETT. Data at the end of each period was combined for the febuxostat and the placebo arms
Time Frame: At the end of each 6 week treatment period (Week 6 and Week 12)
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug, with ischemic chest pain.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 0 | 1
seconds |  | 330 (NA) — Standard deviation cannot be calculated for 1 participant.

11. Secondary Outcome: Exercise Duration
Description: Exercise duration is the exercise time in seconds during ETT. Data at the end of each period was combined for the febuxostat and the placebo arms.
Time Frame: At the end of each 6 week treatment period (Week 6 and Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 30 | 28
seconds | 702 [682.1 to 721.6] | 722 [700.5 to 742.9]

ADVERSE EVENTS:
Time Frame: First dose of study drug to up to 30 days after the last dose of study drug (Up to 16 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Febuxostat 80 mg
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 7/30 | 6/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Febuxostat 80 mg (N=30)
Common cold (Infections and infestations) | 3 | 1
Headache (Nervous system disorders) | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.